CLINICAL TRIAL: NCT05278468
Title: Association Between Periodontitis and Coronavirus Disease (COVID-19) On A Sample of Adult Egyptian Patients: A Case Control Study
Brief Title: Association Between Periodontitis and Coronavirus Disease (COVID-19)
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Khaled Gamil Moussa Megahed, principal investigator, Cairo University
Other Study IDs: 24081992
Record Dates: First submitted 2022-03-11; First posted 2022-03-14 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: Adult Egyptian participants attending the diagnostic center at faculty of Dentistry, Cairo University who had positive real-time reverse transcription polymerase chain reaction results for severe acute respiratory syndrome coronavirus-19 (COVID-19) infection.
  Interventions: Other: PCR test for covid-19
- control group: Adult Egyptian participants attending the diagnostic center at faculty of Dentistry, Cairo University with negative positive real-time reverse transcription polymerase chain reaction results for severe acute respiratory syndrome coronavirus-19 (COVID-19) infection.
  Interventions: Other: PCR test for covid-19

INTERVENTIONS:
Other: PCR test for covid-19 — real-time reverse transcription polymerase chain reaction results for severe acute respiratory syndrome coronavirus-19 (COVID-19) infection.

SUMMARY:
The study is a case control study investigating the association between Periodontitis and Coronavirus disease (COVID-19) in Egyptian dental patients attending the oral diagnosis clinic at faculty of Dentistry, Cairo University.

DETAILED DESCRIPTION:
The coronavirus disease of 2019 (COVID-19) has become a new global issue since its outbreak in Wuhan, China, and has claimed millions of lives as a result. Despite having a low fatality rate of 2.1 percent (WHO), the disease has imposed an unacceptable cost on the world due to its high transmissibility and associated morbidity. The causal virus, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), affects not only the respiratory system but also the cerebrovascular system and other important organs

Coronavirus is a highly contagious single-stranded RNA virus that causes mild to severe respiratory infections in humans and animals. SARS-CoV-2, a novel strand of the -coronavirus family, was discovered in Wuhan, China, in late 2019 which spread fast over the world, forcing WHO to designate the disease a global pandemic on March 11, 2020

The SARS-CoV-2 virus infects host cells by adhering to S-protein, a viral transmembrane spike (S) glycoprotein that clings to human cells by binding to angiotensin converting enzyme II (ACE2), a membrane protein that acts as a virus receptor (Walls et al., 2020). To enable viral fusion into target cells, host proteases such as TMPRSS2, cathepsin L, or proprotein convertase furin proteolytically break the S-protein after it binds to ACE2 . SARS-CoV-2 can also boost the expression of ACE2, making it easier for the virus to invade host cells.

Periodontal disease has been proved to be the most common oral condition of human population . It was widely spread in both the developed and developing countries. High prevalence of periodontal disease has been found in adolescents, adults, and older individuals. Smoking, poor oral hygiene, diabetes, medication, age, hereditary and stress were all considered to be the risk factors of periodontal diseases. Overall, they affected about 20-50% of the population around the globe

Gingivitis and Periodontitis are the most common forms of human periodontal diseases. Inflammation of the gingiva is called gingivitis. The gingiva includes all soft tissue surrounding the tooth coronal to the crest of alveolar bone and to a varying extent lateral to the bone, extending to the mucogingival junction. While, the periodontium includes cementum, periodontal ligament, alveolar bone and the gingiva. Periodontitis includes loss of attachment of periodontal tissues from the tooth together with net loss of alveolar bone height. That's why Gingivitis was found to be reversible, while regeneration after the periodontitis destruction was not predictably achievable . The prevalence of periodontitis has been reported by the World Health Organization (WHO) which showed a prevalence of severe periodontitis in around 8-10% of the Population.

Staging was primarily based on presentation of disease severity as well as disease management sophistication. While the grading offered details about the disease's biological characteristics, including a history-based overview of disease progression risk. This classification also assessed the risk of further development of the disease or any potential negative treatment outcomes and how the disease or its treatment could adversely affect the patient's overall health.

Tonetti stated that staging includes four categories (stages I through IV) and is determined by taking into account several variables, including CAL, amount and percentage of bone loss, PD, existence and degree of angular bony defects, involvement of furcation, mobility of the tooth and loss of the tooth due to periodontitis. On this basis, stage I means initial periodontitis, stage II means moderate periodontitis, stage III means severe periodontitis with potential for additional tooth loss while stage IV means severe periodontitis with potential for loss of dentition. Therefore, data on tooth loss, that can be specifically attributed to periodontitis might alter the concept of the stage.

A periodontitis stage I is characterized by interdental CAL from 1 to 2 mm, radiographic bone loss in the coronal third < 15%, PD ≤ 4 mm and mostly horizontal bone loss, however no tooth loss due to periodontitis is detected at this stage. While, a periodontitis stage II case is characterized by interdental CAL from 3 to 4 mm, radiographic bone loss in the coronal third from 15% to 33%, PD ≤ 5mm and mostly horizontal bone loss, however no tooth loss due to periodontitis is detected at this stage. On the other hand, stages III & IV are characterized by interdental CAL ≥ 5 mm and radiographic bone loss extending to the middle or apical third of the root. In stage III, four teeth or less are lost due to periodontitis while in stage IV, five teeth or more are lost due to periodontitis. In addition to stage II complexity, Stage III is characterized by PD ≥ 6 mm, vertical bone loss ≥ 3mm, furcation involvement class II or III and moderate ridge defect. In addition to stage III complexity, stage IV is characterized by severe ridge defect, bite collapse with drifting and flaring of teeth

The immune system and the inflammatory response to these disorders could be a relationship between periodontitis and COVID-19 severity. The synergy between severe COVID-19 and periodontal disease has been theorised to be the outcome of their immunological activation . In 2021 Hu stated that exaggerated immune responses, such as cytokine storm, which is a prevalent pathway in many inflammatory illnesses, are also identified as one of COVID-19's key tissue-damaging mechanisms. COVID-19 and periodontal diseases have similar proinflammatory cytokine production and influence systemic health, according to research.

Periodontal pockets have the potential to function as viral reservoirs. From pockets of severe periodontitis (Stage 3 and 4) patients, herpes simplex virus (HSV), active human cytomegalovirus (HCMV), and other viral species have been discovered. they theorised that periodontal pockets could act as a reservoir for SARS-CoV-2, increasing viral burden in affected people.

Severe systemic inflammation and thrombotic lesions are the main causes of COVID-19 consequences such acute respiratory distress syndrome and multiorgan failure These issues are linked to a number of risk factors and diseases, many of which are also linked to periodontitis. These links between periodontitis and COVID-19 complications could be due to a direct effect of periodontitis on systemic inflammation, an indirect effect of periodontitis on other COVID-19 risk factors, or predisposing conditions that are common to both periodontitis and COVID-19, such as diabetes and genetic variants

Since the beginning of the pandemic, several investigations have supported the link between COVID-19 and periodontal disorders. Increased gingival bleeding was reported in three case reports among COVID-19 patients. After the viral infection stopped, this condition improved clinically . However, these findings were insufficient to establish a link between periodontitis and COVID-19, especially as individuals with COVID-19 are more inclined to ignore dental hygiene when their health is impacted by COVID-19 symptoms. In fact, patients with COVID-19 have higher oral plaque ratings and gingival edema than their matched SARS-CoV 2 negative controls, according to a recent study made by Anand in 2021. This link between COVID-19 and periodontitis does not imply causation, but it does suggest that more research is needed The study aims at determining whether periodontitis and poor oral hygiene are associated with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years old and above.
2. Patient consulting in the outpatient clinic
3. Provide informed consent.

Exclusion Criteria:

1. Patients having problem in opening their mouth or undergoing intermaxillary fixation where oral examination will not be possible.
2. Patients diagnosed with psychiatric problems or intoxicated with alcohol or drugs.
3. Completely edentulous patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients visiting the dedicated COVID Outpatient Clinic who will undergo real-time reverse transcription polymerase chain reaction (rRT-PCR) for the diagnosis of COVID-19 will be recruited for the study. Subsequently, prior to data analysis, the patients for whom complete set of data will be available will be categorized as either case or control depending on the results of rRT-PCR test by the supervisor. Patients who will have positive rRT-PCR results will be included in the case group, and patients with negative results will be included in the control group. Patients in the control group will be scheduled for an oral examination after the negative rRT-PCR, and patients who were positive for the virus (case group) will be scheduled for an oral examination after the completion of treatment when they will be determined to be disease free through a negative rRT-PCR. peridontal examination will be performed.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
The association between Poor oral hygiene and Coronavirus disease (COVID-19). | 1 year
  after periodontal examination to the 2 groups who are subjected to PCR tests, will we find association between them

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Khaled Gamil, Giza, Egypt